CLINICAL TRIAL: NCT00000654
Title: The Tolerance of HIV-Infected Patients With Herpes Group Virus Infections to Oral Doses of FIAU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Oclassen Pharmaceuticals (Industry)
Purpose: Treatment
Other Study IDs: ACTG 122 FIAU; R90-001-01, 02, 03, 04
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Herpes Simplex; HIV Infections; Hepatitis B
Keywords: AIDS-Related Opportunistic Infections; Pyrimidine Nucleosides; Herpesviridae Infections; Drug Evaluation; Antiviral Agents; Hepatitis B
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Hepatitis B; AIDS-Related Opportunistic Infections; Herpesviridae Infections | interventions — fialuridine

INTERVENTIONS:
Drug: Fialuridine

SUMMARY:
To determine the tolerance of HIV-infected patients to TID oral doses of FIAU syrup at 4 different dose levels. To determine the peak and trough blood levels of FIAU and its metabolites during two weeks of oral dosing with FIAU.

The pyrimidine nucleoside analog FIAC and its primary deaminated uracil metabolite FIAU are highly and specifically active compounds in vitro against several herpes group viruses, particularly herpes simplex virus (HSV) types 1 and 2, varicella zoster (VZV), and cytomegalovirus (CMV), as well as hepatitis B virus (HBV). Since FIAU is the primary metabolite of FIAC and the administration of FIAU simplifies the metabolism of FIAC, it is anticipated from clinical studies of FIAC that FIAU will be tolerated at least as well as FIAC. A single-dose, pharmacokinetic (blood level) study showed that FIAC, when taken orally, is readily absorbed into the bloodstream, and most of it is converted to FIAU. Daily oral doses are expected to provide concentrations of FIAU exceeding the in vitro minimum inhibitory concentration for nearly all the herpes group viruses.

DETAILED DESCRIPTION:
The pyrimidine nucleoside analog FIAC and its primary deaminated uracil metabolite FIAU are highly and specifically active compounds in vitro against several herpes group viruses, particularly herpes simplex virus (HSV) types 1 and 2, varicella zoster (VZV), and cytomegalovirus (CMV), as well as hepatitis B virus (HBV). Since FIAU is the primary metabolite of FIAC and the administration of FIAU simplifies the metabolism of FIAC, it is anticipated from clinical studies of FIAC that FIAU will be tolerated at least as well as FIAC. A single-dose, pharmacokinetic (blood level) study showed that FIAC, when taken orally, is readily absorbed into the bloodstream, and most of it is converted to FIAU. Daily oral doses are expected to provide concentrations of FIAU exceeding the in vitro minimum inhibitory concentration for nearly all the herpes group viruses.

HIV-infected patients with Karnofsky scores at least 80 (with or without documented recurrent herpes group infections) are successively entered into consecutively studied, escalating dose cohorts. There are a total of 4 dose cohorts of FIAU and each patient takes the required amount of FIAU syrup every 8 hours, 1 hour prior to or 3 hours after meals, for a total of 14 days. Entry of new patients at the next higher dose is based on results of tolerance and safety data for prior cohort when all 10 have received 14 days of therapy and at least 7 have met all of the tolerance criteria. Although not formally randomized due to the sequential nature of the study and serious medical condition of the patients, every attempt to avoid bias in assigning a patient to a dose is made. Patients are entered starting with the first dose cohort. Upon meeting the enrollment and tolerance criteria for dose escalation, up to 5 patients with a history of chronic HBV infection and surface antigen positive at their screening visit are added to the end of each dose cohort. Plasma samples are taken to determine peak and trough levels of FIAU at Days 1, 3, 7, and 14 or at last visit. Patients with ongoing active infections are followed by culture (HSV, VZV and CMV) or test (HBV) at Days 1, 3, 7, and 14. Antiemetic therapy with Reglan, Compazine, and Trilafon is given concomitantly at the discretion of the investigator and tolerance determined with antiemetic therapy ongoing. Patients are advised to avoid heavy exercise within 24 hours of any laboratory tests.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Pentamidine aerosol for prophylaxis of recurrent Pneumocystis carinii pneumonia (PCP) in patients currently receiving such treatment.
* Zidovudine (AZT).

Prior Medication:

Allowed:

* Zidovudine (AZT) but only if patient has been taking the drug for > 6 weeks at a dose = or < 600 mg/day, and had < 10 percent decrease in hematocrit, neutrophils, and platelets in the last 30 days.

Patients must:

* Have a diagnosis of HIV infection by ELISA or Western blot. Be able to participate as an outpatient.
* Be ambulatory.
* Have Grade 0 or 1 AIDS Clinical Trial Group toxicity grades for specified laboratory tests.
* Be competent to sign informed consent.
* Be able to cooperate with the treatment plan and evaluation schedule.

NOTE:

* The screening tests must be initiated and completed within 4 weeks prior to the first dose of FIAU, except for diagnostic herpes simplex virus (HSV), varicella zoster (VZV), or cytomegalovirus (CMV) cultures which may have been done previously.
* Concomitant diseases allowed:
* Stable mucocutaneous disease.
* Superficial or uncomplicated infections such as thrush.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* HIV wasting syndrome (involuntary weight loss > 10 percent of baseline body weight and/or chronic diarrhea or weakness and documented fever for at least 30 days).
* Clinical or x-ray evidence of bronchitis, pneumonitis, pulmonary edema, effusion, or suspected active tuberculosis.
* Any unstable medical condition including serious infections or cardiovascular, oncologic, renal, or hepatic condition.
* Primary or initial infection with herpes simplex (HSV), varicella zoster (VZV), or hepatitis B (HBV).
* Cytomegalovirus (CMV) end organ disease.
* Kaposi's sarcoma requiring chemotherapy.
* Systemic fungal infection requiring amphotericin therapy.
* Diagnosis of idiopathic thrombocytopenic purpura (persistent platelet counts < 100000 platelets/mm3 for = or > 3 months).

Patients with the following are excluded:

* HIV wasting syndrome.
* Clinical or x-ray evidence of bronchitis, pneumonitis, pulmonary edema, effusion, or suspected active tuberculosis.
* Any unstable medical condition including serious cardiovascular, infections, oncologic, renal, or hepatic condition.
* Primary or initial infection with herpes simplex (HSV), varicella zoster (VZV), or hepatitis B (HBV).
* Cytomegalovirus (CMV) end organ disease.

Prior Medication:

Excluded within 4 weeks of study entry:

* Ganciclovir (DHPG).
* Foscarnet.
* Interferon.
* Other drug with putative antiviral activity (except zidovudine (AZT)).
* Any immunostimulating drug not specifically allowed.

Excluded within 1 week of study entry:

* Acyclovir.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78
Dates: Study Completion 1993-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D Richman, Study Chair
Locations (4):
- United States (4):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Natl Institute of Health, Bethesda, Maryland
  - Univ of Washington / Madison Clinic, Seattle, Washington

REFERENCES:
- [Background] Tartaglione T, Hooton TM, Jones T, Smiles K, Corey L. Actg 122: phase II tolerance study of oral FIAU in HIV-infected persons. Int Conf AIDS. 1991 Jun 16-21;7(2):254 (abstract no WB2290)